CLINICAL TRIAL: NCT01218347
Title: Influence of OATP1B1 Genotype on the Pharmacokinetics,Lipid Lowering Effect, and Lipid Profiles After Rosuvastatin Administration
Brief Title: Influence of Organic Anion Transporting Polypeptide1B1(OATP1B1) Genotype on Rosuvastatin PK, PD and Lipid Profiles
Acronym: OATP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Kyung-Sang Yu/Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCPT10_Rosuvastatin_OATP1B1
Record Dates: First submitted 2010-10-04; First posted 2010-10-11 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Organic Anion Transporting Polypeptide1B1 (OATP1B1); Rosuvastatin
Keywords: OATP1B1; rosuvastatin
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin (Experimental): rosuvastatin treatment
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 20 mg once daily for 21 days

SUMMARY:
This study aimed to explore the influence of organic anion transporting polypeptide1B1 (OATP1B1) genotype on pharmacokinetics, lipid lowering effect and lipid profiles after rosuvastatin administration.

DETAILED DESCRIPTION:
Open, one arm, single sequence study for healthy volunteers are investigated. Thirty four subjects may be enrolled.

Rosuvastatin are administered once a day for 21 days. Before and after rosuvastatin administration, PK, PD and lipid profiles are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20 to 50 years of age, inclusive (age based on the date to give the informed consent)
* Weight: Over 55 kg, within ±20% of ideal body weight
* Must be reliable and willing to make themselves available during the study period
* Must be willing to give blood sample for genotyping

Exclusion Criteria:

* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease
* History of a significant surgical resection of gastrointestinal tract except appendectomy
* History or evidence of drug abuse
* Use any medication during the last 14 days period before first dosing
* Hypersensitivity to HMG-CoA reductase inhibitor
* Judged to be inappropriate for the study by the investigator

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters(Tmax,Cmax,AUC) of rosuvastatin | Day 21 0h, 1h, 2h, 3h, 4h, 5h, 8h, 12h, 24h

SECONDARY OUTCOMES:
lipid panel(LDL,HDL,TG,Total cholesterol) | Day 1 0h, Day 22 0h
lipid metabolites | Day -1 0h, Day21 0h, 4h, 8h

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University College of Medicine and Hospital
Locations (1):
- Clinical Trials Center, Seoul National University Hospital, Seoul, South Korea